CLINICAL TRIAL: NCT01460264
Title: BIG3 - An Open Prospective Longitudinal Pulmonary-cardiovascular Cohort Study
Brief Title: An Open Prospective Longitudinal Pulmonary-cardiovascular Cohort Study
Acronym: BIG3
Status: Enrolling by invitation | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: BIG3-Region_Skane
Record Dates: First submitted 2011-10-25; First posted 2011-10-26 (Estimated); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Cardiovascular Diseases; Lung Cancer
Keywords: Prospective Cohort Study; Respiratory Function Tests; Computed Tomography; Electrocardiography; Peripheral Arterial Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cardiovascular Diseases; Lung Neoplasms; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- exposed: current daily smokers 100 cigarettes or more during lifetime
- unexposed: current non-smokers

SUMMARY:
This is an observational study aiming to identify and validate biomarkers (including imaging and clinical descriptors) for chronic obstructive pulmonary disease (COPD), cardiovascular disease (CVD) and lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* 45-75 years

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample,residents in Skåne county Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2013-10-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Louise Hagman Bennet, MD, PhD, Study Chair — Skane University Hospital; David Erlinge, MD, PhD, Principal Investigator — Skane University Hospital; Claes-Göran Löfdahl, MD, PhD, Principal Investigator — Skane University Hospital; Maria Planck, MD, PhD, Principal Investigator — Skane University Hospital
Locations (1):
- Skåne University Hospital, Lund, Sweden

REFERENCES:
- [Background] Gerhardsson de Verdier M. The big three concept: a way to tackle the health care crisis? Proc Am Thorac Soc. 2008 Dec 1;5(8):800-5. doi: 10.1513/pats.200806-058TH. PMID 19017732